CLINICAL TRIAL: NCT03690778
Title: A Randomized, Open-label, Single Dose, Crossover Study to Compare the Pharmacokinetic Characteristics of the Co-administration of Metformin SR and Rosuvastatin and JLP-1310 (1000/10mg) in Healthy Male Volunteers.
Brief Title: The PK Characteristics of the Co-administration of Metformin SR and Rosuvastatin and JLP-1310 in Healthy Male Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: JLP-1310-104-PK
Record Dates: First submitted 2018-09-27; First posted 2018-10-01 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Diabetes; Hyperlipidemias
MeSH Terms: conditions — Diabetes Mellitus; Hyperlipidemias | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): Period I: administration of "Metformin" and "Rosuvastatin" seperately Period II: JLP-1310
  Interventions: Drug: "Metformin" and "Rosuvastatin" seperately; Drug: JLP-1310
- Group II (Experimental): Period I: JLP-1301 Period II: administration of "Metformin' and "Rosuvastatin" seperately
  Interventions: Drug: "Metformin" and "Rosuvastatin" seperately; Drug: JLP-1310

INTERVENTIONS:
Drug: "Metformin" and "Rosuvastatin" seperately — administration of "Metformin" and "Rosuvastatin" seperately
Drug: JLP-1310 — administration of JLP-1310

SUMMARY:
A randomized, open-label, single dose, crossover study to compare the pharmacokinetic characteristics of the co-administration of metformin SR and rosuvastatin and JLP-1310 in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteer, age is over 19 years Body weight is over 50 kg, The result of Body Mass Index(BMI) is not less than 18.0 kg/m2 , no more than 29.0 kg/m2.
* Subject who has the ability to comprehend the study objectives, contents and the property of the study drug before participating in the trial.
* Subject who has the ability and willingness to participate the whole period of trial.

Exclusion Criteria:

* Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in kidney, liver, cardiovascular system, respiratory system, endocrine system, or neuropsychiatric system.
* Subjects who are allergic to investigational drug.
* Subjects who have a medical history which can affect the clinical trial.
* 100 mmHg ≥ Systolic BP ≥ 150mmHg or 55 mmHg ≥ Diastolic BP ≥ 95 mmHg
* AST or ALT > X 2 UNL
* Total bilirubin > 2.0 mg/dL
* CK > X 2 UNL
* eGFR < 60 mL/min/1.73m2
* History of drug abuse or positive drug screening.
* Participation in other drug studies within 3 months prior to the drug administration.
* Whole blood donation within 60 days, blood component donation within 30 days or who got transfusion within 30days.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
AUCt of Metformin and rosuvastatin | 48 hours
Cmax of Metformin and rosuvastatin | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Inha University Hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No